CLINICAL TRIAL: NCT06642818
Title: Evaluation of the Effectiveness of PREVENIR (PREVention ENvIronnement Reproduction) Platforms on Urinary Markers of Chemical Exposures - Unblinded Randomized Clinical Trial. PREVENIR-G
Brief Title: Evaluation of the Effectiveness of PREVENIR (PREVention ENvIronnement Reproduction) Platforms
Acronym: PREVENIR-G
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/21
Record Dates: First submitted 2024-04-10; First posted 2024-10-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy; Environmental Exposure; Prevention
Keywords: Pregnancy; Environmental exposure; Prevention

STUDY DESIGN:
Intervention Model Description: Unblinded randomized clinical superiority trial in two parallel groups (intervention vs. no intervention) national multicentre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): During the inclusion visit, urine collection jars will be given to the patient for collection at inclusion and at 3 months. Within the week after the inclusion visit: urine collection will be performed twice a day during 3 days at the patient's home and will be stored in the refrigerator at the participants' home. In the week following this collection, the PREVENIR platforms will be used. At three months, the clinical research officer will contact the patient to remind her of the need to collect urine twice a day during 3 days. This urine collection will be carried out with the same organization as at inclusion. Then, after this urine collection, all the participating women will be interviewed, with a questionnaire identical to the one used for the face-to-face inclusion, in order to allow for the measurement of exhaled Carbon Monoxide (CO). Within 3 to 5 months after inclusion, participating women of the intervention group only,will be invited to participate to the qualitative study.
  Interventions: Other: protocolized interview and prevention messages
- Non-intervention group (No Intervention): During the inclusion visit, urine collection jars will be given to the patient for collection at inclusion and at 3 months. Within the week after the inclusion visit: urine collection will be performed twice a day during 3 days at the patient's home and will be stored in the refrigerator at the participants' home. At three months, the clinical research officer will contact the patient to remind her of the need to collect urine twice a day during 3 days. This urine collection will be carried out with the same organization as at inclusion. Then, after this urine collection, all the participating women will be interviewed, with a questionnaire identical to the one used for the face-to-face inclusion, in order to allow for the measurement of exhaled CO. In the non-intervention group, the full intervention will take place at this time. The control group is a waiting list type control group. The procedure will be performed at the end of the study, i.e. three months after inclusion.

INTERVENTIONS:
Other: protocolized interview and prevention messages — This care consists of a consultation carried out by an environmental health expert (midwife, environmental health engineer) from the PREVENIR platforms. This consultation is carried out through a protocolized interview already developed which allows the identification of exposure to risk factors on reproduction. During the interview, prevention messages targeted at the exposures identified during the interview are delivered.
  Arms: Intervention group

SUMMARY:
Unblinded randomized clinical superiority trial in two parallel groups (intervention vs. no intervention) national multicentre to evaluate the effectiveness of the platforms on the evolution of phenoxyacetic acid levels measured in the urine at inclusion and 3 months after the intervention for patients who received the intervention compared to patients who did not receive the intervention.

DETAILED DESCRIPTION:
it is now recognized that there is a link between certain environmental exposures (occupational and extra-occupational) and reproductive pathologies. During pregnancy, environmental exposures are associated with an increased risk of spontaneous miscarriage, congenital malformations, certain adverse outcomes (fetal death in utero, intrauterine growth retardation, prematurity) and could also increase the risk of chronic disease in childhood and adulthood (hypothesis of developmental origins of health and disease), and have transgenerational effects. Intervention studies have shown efficacy in reducing exposures to certain chemicals, particularly by reducing exposure to cosmetics. In the scientific literature, a pre-conception visit is recommended to identify environmental exposures. In France, platforms are dedicated to the evaluation of environmental exposures in patients with fertility disorders and pregnancy-related pathologies and provide support for the implementation of targeted prevention actions.

The intervention is taken care of by the PREVENIR platforms. This care consists of a consultation carried out by an environmental health expert (midwife, environmental health engineer) from the PREVENIR platforms. This consultation is carried out through a protocolized interview already developed which allows the identification of exposure to risk factors on reproduction. During the interview, prevention messages targeted at the exposures identified during the interview are delivered.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women less than 24 SA of age referred to the PREVENIR platforms participating in the study for management.
* Only women less than 24 SA months pregnant will be included to limit the number of women who gave birth during the study.
* More than 18 years old

For qualitative study:

* Professionnal working within PREVENIR platforms
* Women included in the intervention group and who agreed with participating

Exclusion Criteria:

* Women under court protection, under guardianship or curatorship, severely altered physical and/or psychological health, which, in the opinion of the investigator, may affect the participant's compliance to the study.
* Women with an altered medical condition related to prgnancy that may required a therapeutic abortion according to the environmental expert
* Non-French speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Urinary phenoxyacetic acid concentration | 3 months
  Difference in urinary phenoxyacetic acid concentration between inclusion and 3 months after the intervention. This difference will be compared between the group that received the intervention and the group that did not.

SECONDARY OUTCOMES:
Urinary levels of pyrethroids | 3 months
  Difference in urinary levels of pyrethroids between the intervention and non-intervention groups between baseline and 3 months post intervention
Occupational exposures characterization | 3 months
  During the patient interview, participants will be asked about their occupation, the sector of activity of their employer, the company's size and location, as well as their tasks and the tasks of nearby colleagues. The responses will be analyzed by the environmental health expert conducting the interview, enabling the assessment of occupational exposure to reproductive risk factors in terms of probability, frequency, and intensity.
Chemical exposome | 3 month
  Difference in concentration in urine of chemicals identified by a non-targeted analytical approach (method of analysis without prior knowledge of the substances to be identified)
Endogenous metabolome | 3 months
  Difference in concentration in urine of metabolite identified by a non-targeted analytical approach (method of analysis without prior knowledge of the substances to be identified)
Exhaled CO concentration | 3 months
  Exhaled CO concentration in air between the intervention and non-intervention groups at 3 months post-intervention
Urinary phenoxyacetic acid concentration | 3 months
  Urinary phenoxyacetic acid concentration described according to socio-professional categories
Transferability of the intervention | 5 months
  It will be assessed by examining the dimensions of reach, effectiveness, adoption, implementation and sustainability. It will be measured using a qualitative approach through interviews of professionals and patients. To assess transferability based on validated criteria, we will draw upon established frameworks such as RE-AIM, PARiHS, and TIDieR, which consider multiple factors: relevance to other contexts, local feasibility, social acceptability, and adaptability without loss of effectiveness. The aim is to generate evidence-based recommendations regarding the adaptations required for implementation in alternative settings, to identify the minimum enabling conditions for successful transfer, and to highlight critical factors likely to be sensitive to contextual variation. Conducting the qualitative study across diverse platforms and territorial settings will provide a nuanced understanding of how contextual differences shape implementation processes and outcomes.
Professionals' perceptions | 5 months
  Professional perceptions and practices regarding the prevention of environmental exposures will be explored through semi-structured interviews with professionals working within the PREVENIR platforms. The interview guide will be structured around several thematic areas: representations of environmental risks, preventive practices implemented, perceived barriers and facilitators, and the implicit norms shaping action within the platforms. An inductive thematic analysis will be conducted to identify professional and organizational dynamics that may influence the effectiveness of the platforms in the field of environmental exposure prevention
Professionals' and patients' appreciation and perceived effectiveness | 5 months
  The appreciation and perceived effectiveness of the intervention will be explored through semi-structured interviews with professionals and patients. For professionals, the interview guide will cover themes such as their perception of the intervention, its relevance to professional practice, satisfaction with resources and processes, observed impacts in patient follow-up, as well as barriers and facilitators to its implementation within the platforms. For patients, the themes will include understanding of the intervention, lived experience, satisfaction with the support received, perceived impacts on daily life, appropriation of preventive messages, and barriers and suggestions for improvement. An inductive thematic analysis will be conducted to identify key dimensions influencing satisfaction and perceived effectiveness, as well as factors facilitating or hindering the appropriation of the intervention.
Determinants influencing patients' engagement | 5 months
  The determinants influencing patient engagement in the intervention will be explored through semi-structured interviews. The interview guide will address barriers and facilitators to adherence to recommended measures, as well as the nature and extent of behavioral changes related to environmental exposures. Patients' experiences and perceptions will be collected to identify key facilitators and obstacles to effective participation. An inductive thematic analysis will be conducted to illuminate the underlying dynamics that promote or hinder adherence and behavioral modifications within the context of environmental exposure prevention.
Implementation-related factors | 5 months
  Implementation-related factors will be explored through semi-structured interviews incorporating a set of factual questions designed to collect precise data on the context of consultations. These questions will focus on aspects such as the average duration of consultations, the profession of participants, the possible presence of a partner during the interviews, among others. This collection of factual information will be complemented by open-ended questions to deepen the understanding of organizational and relational conditions influencing implementation. The interviews will be analyzed using an inductive thematic approach to highlight the dynamics and constraints associated with these factors.
Proportion of individuals exposed to occupational reproductive risk factors | 3 months
  Proportion of individuals exposed to occupational reproductive risk factors at 3 months, comparing the intervention and control groups
Urinary levels of parabens | 3 months
  Difference in urinary levels of parabens between the intervention and control groups from baseline to 3 months post-intervention
Urinary levels of phthalates | 3 months
  Difference in urinary levels of phthalates between the intervention and control groups from baseline to 3 months post-intervention
Urinary levels of bisphenols | 3 months
  Difference in urinary levels of bisphenols between the intervention and control groups from baseline to 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fleur DELVA, MD, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delva F, Sentilhes L, Francis-Oliviero F, Bessonneau V, Sunyach C, Audouin C, Paris C, Haddad B, Matrat M, Pairon JC, Belacel M, Sitta R, Roberts T, Bretelle F, Garlantezec R. Evaluation of the efficacy of PREVENIR (PREVention ENvIronment Reproduction) platforms on urinary markers of chemical exposure in pregnant women: protocol for an unblinded randomised clinical trial (PREVENIR-G). BMJ Open. 2025 Nov 9;15(11):e097795. doi: 10.1136/bmjopen-2024-097795. PMID 41213668